CLINICAL TRIAL: NCT04220268
Title: Clinical Database and Biobank of Pulmonary Ground Glass Nodules Patients With Family History, a Prospective Cohort Study.
Brief Title: A Prospective Cohort of Pulmonary Ground Glass Nodules Patients With Family History.
Acronym: GGN-F
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Wen-zhao ZHONG, Porfessor, Guangdong Provincial People's Hospital
Other Study IDs: GGN-family
Record Dates: First submitted 2020-01-05; First posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Lung Neoplasms; Family Research
Keywords: Ground glass nodule; Family aggregation; Hereditary susceptibility
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood and surgical tumor samples of all the participants will be collected. Moreover, blood samples of other family members of participants will be collected, with their consent and knowledge.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: All the patients with proved malignant ground glass nodule will be enrolled.

SUMMARY:
The aim of the present prospective cohort study (GGN-F) is to study the family aggregation of pulmonary ground glass nodules via the questionnaire survey and to investigate the underlying genetic mechanism via the biobank.

DETAILED DESCRIPTION:
In recent years, with the development of low-dose chest CT screening, more and more ground glass nodules have been found. Meanwhile, presenting as Ground-glass nodule (GGN), the early-stage lung adenocarcinoma patients with lung cancer family history have been emerging increasing in recent years in East Asian.

This prospective cohort study, with both a cross-sectional and a longitudinal part, will include patients with pulmonary ground glass nodule, which were proven malignant disease.

All participants will be asked to complete questionnaire to build the clinical database of GGN patients with detailed family history. Furthermore, blood and surgical tumor samples will be collected as a specific biobank. And the blood samples of other family members of participants will be collected, with their consent and knowledge.

ELIGIBILITY:
Inclusion Criteria:

1. patients with informed consent;
2. patients with pulmonary ground glass nodule.
3. pathological proved early stage lung cancer.

Exclusion Criteria:

1.not included in the inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients with pulmonary ground glass nodules and pathological proved malignant disease will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-01-05 (Actual); Primary Completion 2022-01-05 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
The prevalence of family aggregation of pulmonary ground glass nodule. | 1 week
  To investigate the aggregation of pulmonary ground glass nodule among first-degree relatives of participants via the questionnaire.

SECONDARY OUTCOMES:
Susceptibility genetic events related to the family aggregation of ground glass nodules. | 1 month
  To investigate the underlying susceptibility genetic loci which concern with familial inheritance of ground glass nodule.

CONTACTS AND LOCATIONS:
Overall Officials: Wenzhao Zhong, Ph。D, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dai J, Lv J, Zhu M, Wang Y, Qin N, Ma H, He YQ, Zhang R, Tan W, Fan J, Wang T, Zheng H, Sun Q, Wang L, Huang M, Ge Z, Yu C, Guo Y, Wang TM, Wang J, Xu L, Wu W, Chen L, Bian Z, Walters R, Millwood IY, Li XZ, Wang X, Hung RJ, Christiani DC, Chen H, Wang M, Wang C, Jiang Y, Chen K, Chen Z, Jin G, Wu T, Lin D, Hu Z, Amos CI, Wu C, Wei Q, Jia WH, Li L, Shen H. Identification of risk loci and a polygenic risk score for lung cancer: a large-scale prospective cohort study in Chinese populations. Lancet Respir Med. 2019 Oct;7(10):881-891. doi: 10.1016/S2213-2600(19)30144-4. Epub 2019 Jul 17. PMID 31326317